CLINICAL TRIAL: NCT05093465
Title: A Comparison Trial of Two Behavioral Sleep Interventions to Improve Sleep-related Outcomes and Reduce Technology Usage Among College Students
Brief Title: A Comparison of Two Behavioral Sleep Interventions Among College Students (ProjectTECH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oakland University (Other)
Collaborators: Florida State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRBID1306257
Record Dates: First submitted 2021-10-14; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Sleep Disturbance; Sleep Hygiene
MeSH Terms: conditions — Parasomnias; Sleep Hygiene

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Control (Active Comparator): Participants were provided with sleep hygiene and stimulus control procedures.
  Interventions: Other: Active Control
- Technology Intervention (Experimental): Participants were given the same intervention materials as the active control condition plus procedures to change technology use.
  Interventions: Behavioral: Technology Intervention

INTERVENTIONS:
Behavioral: Technology Intervention — Participants were provided with sleep hygiene and stimulus control procedure plus procedures to reduce technology usage in bed (i.e., technology usage stimulus control).
  In addition to the sleep hygiene and stimulus control procedures, participants were also given a set of procedures aimed at changing technology usage behavior at bedtime and throughout the day.
  Arms: Technology Intervention
Other: Active Control — Participants were provided with sleep hygiene and stimulus control procedures.
  Arms: Active Control

SUMMARY:
The study was a randomized controlled trial designed to examine whether augmenting traditional sleep hygiene and stimulus control procedures with technology use reduction stimulus control procedures would produce better sleep and technology usage outcomes.

DETAILED DESCRIPTION:
Sixty college students were randomized to a 4-week sleep hygiene and stimulus control intervention (ACI) or an enhanced intervention including technology stimulus control instructions (TI).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years old, enrolled at Oakland University, and reside in an on-campus dormitory to participate.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | From baseline to posttest, approximately 5 weeks
  Scores on the Pittsburgh Sleep Quality Index
Technology Usage | From baseline to posttest, approximately 5 weeks
  Self-reported usage of various forms of technology in minutes

SECONDARY OUTCOMES:
Sleep Hygiene | From baseline to posttest, approximately 5 weeks
  Scores on the Sleep Hygiene Practice Scale
Sleep Control | From baseline to posttest, approximately 5 weeks
  Scores on the Motivation Survey

CONTACTS AND LOCATIONS:
Overall Officials: Andrea T Kozak, PhD, Principal Investigator — Oakland University
Locations (1):
- Oakland University, Rochester, Michigan, United States

IPD SHARING:
Plan to Share IPD: No